CLINICAL TRIAL: NCT03022643
Title: Social & Behavioral Rhythms in Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Ariel Neikrug, Postdoctoral Fellow, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 094507
Record Dates: First submitted 2016-11-18; First posted 2017-01-16 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Patients (No Intervention): 40 Pain Patients will be screened for social and behavioral rhythms with no treatment involved. All patients will be evaluated an Actigraph by Philips for 8-days to assess sleep and activity.
- Controls (No Intervention): 40 Controls will be screened for social and behavioral rhythms with no treatment involved. All Controls will be evaluated an Actigraph by Philips for 8-days to assess sleep and activity.
- Treatment (Experimental): 10 patients from the original 40 will receive Interpersonal Social Rhythms Psychotherapy and Bright Light Device therapy to improve social and behavioral rhythms.
  Interventions: Behavioral: Interpersonal Social Rhythms Psychotherapy; Other: Bright Light Device

INTERVENTIONS:
Behavioral: Interpersonal Social Rhythms Psychotherapy — The treatment involves 8-weeks of individual psychotherapy. Weekly sessions will be 60-minute long and will take place at the Pain Research Center. The treatment focuses on 1) the link between life events, pain severity, sleep disturbances, fatigue, and mood, 2) social and behavioral rhythms and sleep-wake disturbances, 3) identification and management of rhythm dysregulation and the triggers for it, 4) allowing and facilitating the mourning of the loss healthy self, 5) identification and appropriate management of symptoms.
  Arms: Treatment
Other: Bright Light Device — All patients will be provided with a bright light device (Re-Timer) and will be instructed to use it in the first 2-hours of the day (for a minimum of 30 minutes) throughout the 8-week treatment period.
  Other Names: Re-Timer
  Arms: Treatment

SUMMARY:
Behavioral and biological rhythms are essential for health. No study evaluated behavioral rhythm or rhythm regulation in chronic pain and how this impacts functioning. The objective of this study is to gather preliminary data, focusing on the role of behavioral rhythms in the cardinal clinical symptoms of chronic pain (i.e., sleep, fatigue, and mood). Additionally, this study will provide preliminary data for the feasibility and acceptability of the therapeutic approach aiming to strengthen behavioral rhythms for patients with chronic pain.

DETAILED DESCRIPTION:
The overall goal of this study is to gather preliminary data, focusing on behavioral rhythms in patients with chronic pain as well as the relationship between behavioral rhythms and the pain-related clinical symptoms. Additionally, this study will provide preliminary data for the feasibility, acceptability, and treatment effects of repurposing interpersonal social rhythm therapy (IPSRT) along with light therapy for patients with chronic pain exhibiting significant rhythm dysregulation, sleep disturbances, and mood symptoms. The deliverables at the end of this project will include 1) preliminary evidence concerning the prevalence of behavioral rhythm disturbances in patients with chronic pain; 2) the association between such behavioral rhythm disruptions and the symptom cluster of pain-sleep-fatigue-mood; 3) feasibility and acceptability of a prototype IPSRT repurposed for chronic pain patients along with bright light therapy. The specific aims of this proposed study are as follows:

Aim 1: To evaluate regularity of social and behavioral rhythms (SBR), disruption of circadian activity rhythms (CAR), and the relationship of SBR and CAR with clinical symptoms of pain-sleep-fatigue-mood in chronic pain patients compared to healthy control.

Hypothesis 1: Patients with chronic pain will show high degrees of SBR and CAR disruption compared to controls.

Hypothesis 2: Patients with increasingly dysregulated SBR and attenuated CAR will exhibit worse clinical symptoms.

Hypothesis 3: SBR will be associated with CAR in patients with chronic pain and in controls.

Aim 2: To assess feasibility and acceptance of interpersonal social rhythm therapy repurposed for chronic pain patient population along with bright light therapy provided to patients exhibiting SBR disruption with significant sleep and mood symptoms.

Hypothesis 1: The IPSRT will be well tolerated and accepted by the patients

Hypothesis 2: Descriptive data will suggest improvement of SBR, CAR, and the pain-related symptoms and functioning.

ELIGIBILITY:
Inclusion Criteria:

All participants (patients and controls):

* 18-65 years of age with
* reading/writing proficiency in English.

Aim 1:

Patients must:

* have had persistent pain for more than 1-year at a consistent body part or diffuse body pain (e.g., fibromyalgia) that is stable rather than progressive in nature
* report experiencing pain for more than 70% of the waking hours in any given week
* under current medical care by a physician for a pain diagnosis
* able remain stable on any of their medication (as prescribed) for the duration of the 8-day evaluation involved in Aim 1

Control subjects must:

* be pain-free for the past 1-year
* no prior treatment for a chronic pain condition
* in overall good health

Aim 2:

Patients must:

* have current symptoms of insomnia (Insomnia Severity Index (ISI), ISI>8)
* have depression (Patient Health Questionnaire-9, PHQ-9>10)
* exhibit significant circadian activity rhythm dysregulation during the 8-day evaluation (defined as Amplitude<0.9)

Control subjects must:

* be pain-free for the past 1-year
* no prior treatment for a chronic pain condition
* in overall good health

Exclusion Criteria:

Aim 1:

* patients/controls who underwent surgery in the last 6-months
* shift workers
* dementia
* current drug abuse/dependence
* receiving treatment in methadone clinic
* current cardiac conditions
* untreated sleep apnea
* untreated restless legs syndrome
* neurodegenerative disease
* bipolar disorder
* psychosis
* suicidal ideation
* have changed time-zones in the last 7 days
* experienced a significant life change in the last month (e.g., death in the family, loss of job, traumatic event)

Aim 2:

* patients/controls who underwent surgery in the last 6-months
* shift workers
* dementia
* current drug abuse/dependence
* receiving treatment in methadone clinic
* current cardiac conditions
* untreated sleep apnea
* untreated restless legs syndrome
* neurodegenerative disease
* bipolar disorder
* psychosis
* suicidal ideation
* have changed time-zones in the last 7 days
* experienced a significant life change in the last month (e.g., death in the family, loss of job, traumatic event)
* receiving psychotherapy
* significant photophobia
* chronic migraines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Activity Rhythms - Actigraphy Assessment | Baseline
  Collected continuously for 8 days at baseline
Change in Activity Rhythms - Actigraphy Assessment | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected continuously for 8 days at baseline, at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)

SECONDARY OUTCOMES:
Insomnia Severity index | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected at baseline (prior the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)
Patient Health Questionnaire-9 (PHQ-9) | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected at baseline (prior the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)
Social Rhythms Metric | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected continuously at baseline (during the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)
Sleep Disturbances: Patient Reported Outcome Measurement System (PROMIS) Short-Form Measures for Sleep disturbance | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected at baseline (prior the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)
Sleep-Related Impairment: Patient Reported Outcome Measurement System (PROMIS) Short-Form Measures for sleep related impairment | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected at baseline (prior the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)
Fatigue: Patient Reported Outcome Measurement System (PROMIS) Short-Form Measures for Fatigue | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected at baseline (prior the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)
Depression: Patient Reported Outcome Measurement System (PROMIS) Short-Form Measures for Depression | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected at baseline (prior the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)
Anxiety: Patient Reported Outcome Measurement System (PROMIS) Short-Form Measures for Anxiety | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected at baseline (prior the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)
Pain Behavior: Patient Reported Outcome Measurement System (PROMIS) Short-Form Measures for Pain behavior | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected at baseline (prior the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)
Pain Interference: Patient Reported Outcome Measurement System (PROMIS) Short-Form Measures for pain interference | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected at baseline (prior the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)
Physical Functioning: Patient Reported Outcome Measurement System (PROMIS) Short-Form Measures for physical functioning | Baseline, Pre-treatment (within 2 weeks of Baseline Assessment), Mid-Therapy (4-weeks), Post-treatment (8-weeks)
  Collected at baseline (prior the 8-day assessment), at Pre-treatment for those receiving the therapy (within 2 weeks of Baseline assessment) as well as at mid point of therapy (4-weeks) and post therapy (8-weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel B Neikrug, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No